CLINICAL TRIAL: NCT01353105
Title: Evaluation and Reconditioning of Marginal Lung Donors to Transplantation by ex Vivo Lung Perfusion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: InCor Heart Institute (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Fabio Biscegli Jatene/ Full Professor of Thoracic Surgery - Medical School, University of São Paulo, InCor Heart Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCOR-1232-09
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2010-10

CONDITIONS: Respiratory Tract Diseases
Keywords: cystic fibrosis; chronic obstructive pulmonary disease; pulmonary fibrosis
MeSH Terms: conditions — Respiratory Tract Diseases; Cystic Fibrosis; Pulmonary Disease, Chronic Obstructive; Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ex vivo lung transplantation (Experimental): single-group studies
  Interventions: Procedure: Ex vivo lung transplantation

INTERVENTIONS:
Procedure: Ex vivo lung transplantation — Evaluation and reconditioning of lungs following lung transplantation
  Other Names: Non applicable

SUMMARY:
Only about 15% of the potential candidates for lung donation are considered suitable for transplantation. A new method for ex vivo lung perfusion (EVLP) has been developed and can be used for evaluation and reconditioning of "marginal" and unacceptable lungs. The ´purpose of this study is to analyse the executability and safety of ex vivo lung perfusion pulmonary ex vivo in marginal donors.

DETAILED DESCRIPTION:
Donor Inclusion criteria:

* Age < 55 years-old;
* Smoking history < 20 pack-year;
* Clear chest radiograph;
* Absence of significant chest trauma;
* Absence of purulent secretions and gastric contents at bronchoscopy;
* PaO2 < 300 mm Hg (FIO2 1.0, PEEP 5 cmH2O)

Exclusion criteria:

* Lungs presenting PO2 < 400 mmHg after ex vivo lung perfusion

ELIGIBILITY:
Inclusion Criteria:

* Age < 55 years-old;
* Smoking history < 20 pack-year;
* Clear chest radiograph;
* Absence of significant chest trauma;
* Absence of purulent secretions and gastric contents at bronchoscopy;
* PaO2 < 300 mm Hg (FIO2 1.0, PEEP 5 cmH2O)

Exclusion Criteria:

* Lungs presenting PO2 < 400 mmHg after ex vivo lung perfusion

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
30-days mortality | 30 days after ex vivo lung transplantation
Respiratory complications (primary graft dysfunction, infection, rejection, bronchiolitis obliterates syndrome) | 30 days after the ex vivo lung transplantation
12-months survival | 12 months survival after ex vivo lung transplantation

SECONDARY OUTCOMES:
Oxygenation index (PaO2/FiO2)on ICU arrival and 72 hours | 72 hours after ex vivo lung transplantation
Mechanical ventilation time | 30 days after ex vivo lung transplantation
Hospital and ICU time of stay | 12 months after ex vivo lung transplantation
Non-respiratory complications (arrhythmia, renal failure, sepsis) | 30 days after ex vivo lung transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Fabio B Jatene, PhD, Principal Investigator — InCor Heart Institute
Locations (1):
- INCOR - Heart Institute, São Paulo, São Paulo, Brazil